CLINICAL TRIAL: NCT01819233
Title: A Feasibility Pilot Trial Evaluating Caloric Restriction for Oncology Research in Early Stage Breast Cancer Patients
Brief Title: Caloric Restriction in Treating Patients With Stage 0-I Breast Cancer Undergoing Surgery and Radiation Therapy
Acronym: CAREFOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 12G.616; 2012-94 (Other: CCRRC); JT 3024 (Other: JeffTrial Number); P30CA056036 (NIH)
Record Dates: First submitted 2013-03-22; First posted 2013-03-27 (Estimated); Results first posted 2019-12-23 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Ductal Breast Carcinoma in Situ; Invasive Ductal Breast Carcinoma; Invasive Lobular Breast Carcinoma; Lobular Breast Carcinoma in Situ; Recurrent Breast Cancer; Stage IA Breast Cancer; Stage IB Breast Cancer
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating; Carcinoma, Ductal, Breast; Carcinoma, Lobular; Breast Carcinoma In Situ; Breast Neoplasms | interventions — Radiotherapy; Radiation; Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Behavioral dietary intervention (Experimental): Beginning 2-4 weeks after completion of lumpectomy, patients receive food diaries to complete for 7-10 days. Dietary counselors then give patients guidelines for dietary modifications to reduce caloric intake by 25% of their normal diet. Patients follow caloric restricted diet for 10 weeks (2 weeks prior to radiation therapy, during 6 weeks of radiation therapy, and at least 2 weeks after radiation therapy). Patients undergo radiation therapy QD 5 days a week for 6 weeks.
  Interventions: Behavioral: Behavioral dietary intervention; Procedure: Therapeutic conventional surgery; Radiation: Radiation therapy; Other: Counseling intervention; Procedure: Quality-of-life assessment

INTERVENTIONS:
Behavioral: Behavioral dietary intervention — Receive caloric restricted dietary intervention
Procedure: Therapeutic conventional surgery — Undergo definitive lumpectomy
Radiation: Radiation therapy — Undergo radiation therapy
  Other Names: Irradiation; Radiotherapy; Radiation
Other: Counseling intervention — Receive dietary counseling
  Other Names: Counseling and communications studies
Procedure: Quality-of-life assessment — Ancillary studies
  Other Names: Quality of life assessment

SUMMARY:
This pilot clinical trial studies caloric restriction in patients with stage 0-I breast cancer during surgery and radiation therapy. Reducing caloric intake may prevent disease progression in patients with breast cancer. Radiation therapy uses high energy x rays to kill tumor cells. Giving dietary intervention and radiation therapy together may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

1. Investigate the feasibility of a clinical trial administering ionizing radiation with concurrent caloric restriction (CR) for the treatment of breast cancer.

   SECONDARY OBJECTIVE:
2. Investigate measurable changes of patient characteristics and tissue and serum from CR conditions to determine a metric for evaluating this treatment in future studies.

OUTLINE:

Beginning 2-4 weeks after completion of lumpectomy, patients receive food diaries to complete for 7-10 days. Dietary counselors then give patients guidelines for dietary modifications to reduce caloric intake by 25% of their normal diet. Patients follow caloric restricted diet for 10 weeks (2 weeks prior to radiation therapy, during 6 weeks of radiation therapy, and at least 2 weeks after radiation therapy). Patients undergo radiation therapy once daily (QD) 5 days a week for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically proven diagnosis of ductal carcinoma in situ (DCIS) or invasive breast cancer
2. Ability to have breast conservation as determined by the judgment of the radiation oncologist, for which the radiation oncologist has determined that he or she will only treat the whole breast and not regional lymph nodes
3. The patient must be female
4. Age >= 18
5. If multifocal breast cancer, then it must be able to be resected through a single lumpectomy incision
6. Appropriate stage for protocol entry, including no clinical evidence for distant metastases, based upon the following minimum diagnostic workup:

   1. History/physical examination, including breast exam and documentation of weight and Karnofsky performance status of 80-100% for at least 60 days prior to study entry
   2. Ipsilateral mammogram within 6 months prior to study entry
7. Women of childbearing potential must have a negative serum pregnancy test within 14 days of study entry
8. Women of childbearing potential must be non-pregnant and non-lactating and willing to use medically acceptable form of contraception during radiation therapy
9. Patient must capable of and provide study specific informed consent prior to study entry
10. Body mass index (BMI) >= 21
11. Weight >= 100 lbs
12. No prior history of non-breast malignancies in the past 2 years unless it was a non-melanomatous skin lesion or carcinoma in situ of the cervix
13. Patient must not have any of the following severe, active co-morbidity, defined as follows:

    1. Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months
    2. Transmural myocardial infarction within the last 6 months
    3. Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
    4. Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within 30 days before registration
    5. Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects; note, however, that laboratory tests for liver function and coagulation parameters are not required for entry into this protocol
    6. Acquired immune deficiency syndrome (AIDS) or human immunodeficiency virus (HIV) positive based upon current Centers for Disease and Control (CDC) definition; note, however, that HIV testing is not required for entry into this protocol; the need to exclude patients with AIDS or HIV from this protocol is necessary because anti-retrovirals may alter patient metabolism
14. Patient must not have active systemic lupus, erythematosus, or any history of scleroderma, dermatomyositis with active rash
15. No prior radiotherapy to the ipsilateral breast or prior radiation to the region of the breast that would result in overlap of radiation therapy fields
16. Patient may not have any active gastrointestinal/malabsorption disorder at the discretion of the Principal Investigator

    1. Inflammatory bowel disease
    2. Celiac disease
    3. Chronic pancreatitis
    4. Chronic diarrhea or vomiting
    5. Active eating disorder
17. Creatinine < 1.7
18. Not currently taking steroids
19. No currently active pituitary secreting tumors up to physician discretion
20. No history of or current active drug/alcohol dependence
21. No patients being decisionally impaired

Exclusion Criteria:

1. Patient is not a candidate for breast conservation
2. Patient is male
3. Age < 18 years
4. Patient requires regional lymph node irradiation therapy
5. Patient has evidence of distant metastases
6. Karnofsky performance status less than 80% within 60 days prior to study
7. Ipsilateral mammogram done greater than 6 months prior to study
8. Women of childbearing potential with a positive serum beta human chorionic gonadotropin (hCG)
9. Patient has a history of dementia, psychosis or other disorder affecting their mental status to the point where they cannot consent or comply with study guidelines
10. BMI < 21
11. Weight < 100 lbs
12. Weight loss >= 10% in the last 3 months (mos)
13. Prior invasive non-breast malignancy (except non-melanomatous skin cancer, carcinoma in situ of the cervix) unless disease free for a minimum of 2 years prior to registration
14. Two or more breast cancers not resectable through a single lumpectomy incision
15. Non-epithelial breast malignancies such as sarcoma or lymphoma
16. Prior radiotherapy to the ipsilateral breast or prior radiation to the region of the breast that would result in overlap of radiation therapy fields
17. Severe, active co-morbidity, defined as follows:

    1. Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months
    2. Transmural myocardial infarction within the last 6 months
    3. Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
    4. Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within 30 days before registration
    5. Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects; note, however, that laboratory tests for liver function and coagulation parameters are not required for entry into this protocol
    6. Acquired immune deficiency syndrome (AIDS) or HIV positive based upon current CDC definition; note, however, that HIV testing is not required for entry into this protocol; the need to exclude patients with AIDS or HIV from this protocol is necessary because anti-retrovirals may alter patient metabolism
18. Active systemic lupus, erythematosus, or any history of scleroderma, dermatomyositis with active rash
19. Active gastrointestinal/malabsorption disorder at the discretion of the Principal Investigator

    1. Inflammatory bowel disease
    2. Celiac disease
    3. Chronic pancreatitis
    4. Chronic diarrhea or vomiting
    5. Active eating disorder
20. Creatinine >= 1.7
21. Current use of steroids
22. Pituitary secreting tumors up to physician discretion
23. Active drug/alcohol dependence or abuse history
24. Decisionally impaired patients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2013-03-08 (Actual); Primary Completion 2017-09-14 (Actual); Study Completion 2019-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Simone, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Longo VD, Fontana L. Calorie restriction and cancer prevention: metabolic and molecular mechanisms. Trends Pharmacol Sci. 2010 Feb;31(2):89-98. doi: 10.1016/j.tips.2009.11.004. Epub 2010 Jan 25. PMID 20097433
- [Background] Hursting SD, Lavigne JA, Berrigan D, Perkins SN, Barrett JC. Calorie restriction, aging, and cancer prevention: mechanisms of action and applicability to humans. Annu Rev Med. 2003;54:131-52. doi: 10.1146/annurev.med.54.101601.152156. Epub 2001 Dec 3. PMID 12525670
- [Background] Rous P. THE INFLUENCE OF DIET ON TRANSPLANTED AND SPONTANEOUS MOUSE TUMORS. J Exp Med. 1914 Nov 1;20(5):433-51. doi: 10.1084/jem.20.5.433. PMID 19867833
- [Background] Tannenbaum A. Effects of Varying Caloric Intake Upon Tumor Incidence and Tumor Growth. Annals of the New York Academy of Sciences. 15 Dec 2006 2006;49(1).
- [Background] Berrigan D, Perkins SN, Haines DC, Hursting SD. Adult-onset calorie restriction and fasting delay spontaneous tumorigenesis in p53-deficient mice. Carcinogenesis. 2002 May;23(5):817-22. doi: 10.1093/carcin/23.5.817. PMID 12016155
- [Background] Zhu Z, Jiang W, Thompson HJ. Effect of energy restriction on tissue size regulation during chemically induced mammary carcinogenesis. Carcinogenesis. 1999 Sep;20(9):1721-6. doi: 10.1093/carcin/20.9.1721. PMID 10469616
- [Background] Lok E, Scott FW, Mongeau R, Nera EA, Malcolm S, Clayson DB. Calorie restriction and cellular proliferation in various tissues of the female Swiss Webster mouse. Cancer Lett. 1990 May 15;51(1):67-73. doi: 10.1016/0304-3835(90)90232-m. PMID 2337899
- [Background] Grasl-Kraupp B, Bursch W, Ruttkay-Nedecky B, Wagner A, Lauer B, Schulte-Hermann R. Food restriction eliminates preneoplastic cells through apoptosis and antagonizes carcinogenesis in rat liver. Proc Natl Acad Sci U S A. 1994 Oct 11;91(21):9995-9. doi: 10.1073/pnas.91.21.9995. PMID 7937932
- [Background] Turner BC, Haffty BG, Narayanan L, Yuan J, Havre PA, Gumbs AA, Kaplan L, Burgaud JL, Carter D, Baserga R, Glazer PM. Insulin-like growth factor-I receptor overexpression mediates cellular radioresistance and local breast cancer recurrence after lumpectomy and radiation. Cancer Res. 1997 Aug 1;57(15):3079-83. PMID 9242428
- [Background] Perer ES, Madan AK, Shurin A, Zakris E, Romeguera K, Pang Y, Beech DJ. Insulin-like growth factor I receptor antagonism augments response to chemoradiation therapy in colon cancer cells. J Surg Res. 2000 Nov;94(1):1-5. doi: 10.1006/jsre.2000.5923. PMID 11038295
- [Background] Donohoe CL, Doyle SL, Reynolds JV. Visceral adiposity, insulin resistance and cancer risk. Diabetol Metab Syndr. 2011 Jun 22;3:12. doi: 10.1186/1758-5996-3-12. PMID 21696633
- [Background] Kahn SE, Hull RL, Utzschneider KM. Mechanisms linking obesity to insulin resistance and type 2 diabetes. Nature. 2006 Dec 14;444(7121):840-6. doi: 10.1038/nature05482. PMID 17167471
- [Background] Lee C, Safdie FM, Raffaghello L, Wei M, Madia F, Parrella E, Hwang D, Cohen P, Bianchi G, Longo VD. Reduced levels of IGF-I mediate differential protection of normal and cancer cells in response to fasting and improve chemotherapeutic index. Cancer Res. 2010 Feb 15;70(4):1564-72. doi: 10.1158/0008-5472.CAN-09-3228. Epub 2010 Feb 9. PMID 20145127
- [Background] Safdie F, Brandhorst S, Wei M, Wang W, Lee C, Hwang S, Conti PS, Chen TC, Longo VD. Fasting enhances the response of glioma to chemo- and radiotherapy. PLoS One. 2012;7(9):e44603. doi: 10.1371/journal.pone.0044603. Epub 2012 Sep 11. PMID 22984531
- [Background] National Institutes of Health. http://www.clincaltrials.gov.
- [Background] Arguin H, Dionne IJ, Senechal M, Bouchard DR, Carpentier AC, Ardilouze JL, Tremblay A, Leblanc C, Brochu M. Short- and long-term effects of continuous versus intermittent restrictive diet approaches on body composition and the metabolic profile in overweight and obese postmenopausal women: a pilot study. Menopause. 2012 Aug;19(8):870-6. doi: 10.1097/gme.0b013e318250a287. PMID 22735163
- See also: Kimmel Cancer Center at Thomas Jefferson University, an NCI-Designated Cancer Center — http://www.KimmelCancerCenter.org
- See also: Thomas Jefferson University Hospitals — http://www.JeffersonHospital.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Behavioral Dietary Intervention
Started | 38
Completed | 32
Not Completed | 6

BASELINE CHARACTERISTICS:
Arm/Group | Behavioral Dietary Intervention
Number analyzed (Participants) | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 33
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 33
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 15
  White | 18
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 38

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Are Adherent to the Diet Restriction
Description: Computed along with a 95% exact confidence interval. Exact binomial test (with a one-sided alpha of 0.05) will be used to test whether adherence is greater than 60%.
Time Frame: Up to week 12
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Behavioral Dietary Intervention
Number analyzed (Participants) | 32
participants | 28 [NA to 74.5] — one sided lower confidence limit as one-sided alpha used.

2. Secondary Outcome: Change in Body Fat Measurement
Description: Analyzed via a paired t-test. Change in body fat measurement as determined by the Durnin-Womersley 4-fold technique
Time Frame: Baseline to 4 weeks after completion of study
Population: patients who did not complete all assessments were not included in the analysis
Measure: Mean (95% Confidence Interval); unit: percentage of change in body fat
Arm/Group | Behavioral Dietary Intervention
Number analyzed (Participants) | 29
percentage of change in body fat | -3.1 [-4.7 to -1.5]

3. Secondary Outcome: Change in Body Mass Index (BMI)
Description: Assessed via mixed-effects regression. Weight changes over time assessed by modeling BMI as a function of time
Time Frame: Baseline to 4 weeks after completion of study
Population: participants who did not complete all timepoint measurements were not included.
Measure: Mean (95% Confidence Interval); unit: percentage of change in BMI
Arm/Group | Behavioral Dietary Intervention
Number analyzed (Participants) | 31
percentage of change in BMI | -1.2 [-1.6 to -0.8]

4. Secondary Outcome: Change in Heart Rate Over Time
Description: Assessed via mixed-effects regression.
Time Frame: Baseline to 4 weeks after completion of study
Population: only participants who completed all timepoints were included
Measure: Mean (Standard Error); unit: beats per minute
Arm/Group | Behavioral Dietary Intervention
Number analyzed (Participants) | 32
beats per minute | 67.3 (1.5)

5. Secondary Outcome: Patterns of Change Over Time in Serum Markers
Description: Assessed via mixed-effects regression.
Time Frame: Baseline to 4 weeks after completion of study
Reporting Status: Not Posted

6. Secondary Outcome: Patterns of Change Over Time in Psycho-social Outcomes Measured Using the Functional Assessment of Cancer Therapy-Breast (FACT-B)
Description: Assessed via mixed-effects regression. The FACT-B is a questionnaire using a 5-point Likert scale (0-Not at all to 4-Very much)
Time Frame: Baseline to 4 weeks after completion of study
Population: patients who did not complete all questionnaire timepoints were not included in the analysis
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Behavioral Dietary Intervention
Number analyzed (Participants) | 31
score on a scale | 0.8 [-6.2 to 7.8]

7. Secondary Outcome: Local Recurrence
Description: Analyzed via survival methods, specifically the Kaplan-Meier method and the logrank test.
Time Frame: Up to 4 weeks after completion of study
Measure: Count of Participants; unit: Participants
Arm/Group | Behavioral Dietary Intervention
Number analyzed (Participants) | 38
Participants | NA — Sincere efforts were made to gather and report the data, however, no data is available for this endpoint.

8. Secondary Outcome: Distant Metastases
Description: Analyzed via survival methods, specifically the Kaplan-Meier method and the logrank test.
Time Frame: Up to 4 weeks after completion of study
Measure: Count of Participants; unit: Participants
Arm/Group | Behavioral Dietary Intervention
Number analyzed (Participants) | 38
Participants | NA — Sincere efforts were made to gather and report the data, however, no data is available for this endpoint.

9. Secondary Outcome: Progression Free Survival
Description: Analyzed via survival methods, specifically the Kaplan-Meier method and the logrank test.
Time Frame: Up to 4 weeks after completion of study
Measure: Count of Participants; unit: Participants
Arm/Group | Behavioral Dietary Intervention
Number analyzed (Participants) | 38
Participants | NA — Sincere efforts were made to gather and report the data, however, no data is available for this endpoint.

10. Secondary Outcome: Overall Survival
Description: Analyzed via survival methods, specifically the Kaplan-Meier method and the logrank test.
Time Frame: Up to 4 weeks after completion of study
Population: Insufficient data was collected to conduct survival analysis as there were participants who were lost to follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | Behavioral Dietary Intervention
Number analyzed (Participants) | 38
Participants | NA — Sincere efforts were made to gather and report the data, however, no data is available for this endpoint.

ADVERSE EVENTS:
Time Frame: baseline through 5 weeks after completion of study diet.
Arm/Group | Behavioral Dietary Intervention
All-Cause Mortality (participants affected / at risk) | 0/38
Serious Adverse Events (participants affected / at risk) | 0/38
Other Adverse Events (participants affected / at risk) | 14/38
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Behavioral Dietary Intervention (N=38)
Dermatitis (Skin and subcutaneous tissue disorders) | 13 (38)
fatigue (General disorders) | 13 (38)
hot flashes (General disorders) | 5
hyperpigmentation (Skin and subcutaneous tissue disorders) | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-04): https://cdn.clinicaltrials.gov/large-docs/33/NCT01819233/Prot_SAP_000.pdf